CLINICAL TRIAL: NCT00693108
Title: Transdermal Testosterone to Improve Ovarian Response to Gonadotropins in Poor Responder IVF Patients With Normal Basal Concentrations of FSH
Brief Title: Androgens for Poor Responders in In Vitro Fertilization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Other Study IDs: IVFANDROGENS
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Ovarian Response
Keywords: Poor; Response; Ovarian; Stimulation; IVF; Patients

ARMS (2):
- 1 (Experimental): Transdermal testosterone treatment during the five days preceding gonadotropin therapy in IVF cycles
  Interventions: Drug: Transdermal testosterone
- 2 (No Intervention)

INTERVENTIONS:
Drug: Transdermal testosterone
  Arms: 1

SUMMARY:
it has been shown that androgens in non human primates may favour follicular growth in the ovaries when animals are treated with gonadotropins which are the hormones used in patients receiving treatment with in vitro fertilization. Therefore, this study investigates the potential usefulness of testosterone treatment preceding gonadotropin administration in in vitro fertilization patients having a previous poor response to gonadotropins alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving the second IVF treatment attempt having the first treatment cycle cancelled because of poor ovarian response to gonadotropins

Exclusion Criteria:

* Previous ovarian surgery
* Clinical or laboratory profile suggesting premature ovarian failure

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Background] Balasch J, Fabregues F, Penarrubia J, Carmona F, Casamitjana R, Creus M, Manau D, Casals G, Vanrell JA. Pretreatment with transdermal testosterone may improve ovarian response to gonadotrophins in poor-responder IVF patients with normal basal concentrations of FSH. Hum Reprod. 2006 Jul;21(7):1884-93. doi: 10.1093/humrep/del052. Epub 2006 Mar 3. PMID 16517559